CLINICAL TRIAL: NCT00627692
Title: A Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Tolerability of Oral Once-Daily Prucalopride (R108512) Solution in Constipated Elderly Subjects Living in a Nursing Facility
Brief Title: Evaluation of the Safety and Tolerability of Prucalopride in Constipated Elderly Subjects Living in a Nursing Facility
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Renate Specht Gryp, Movetis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRU-USA-26
Record Dates: First submitted 2008-02-21; First posted 2008-03-03 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-01

CONDITIONS: Constipation
Keywords: Constipation in elderly patients
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Active Comparator): Prucalopride
  Interventions: Drug: Prucalopride
- 2 (Active Comparator): Prucalopride
  Interventions: Drug: Prucalopride
- 3 (Active Comparator): Prucalopride
  Interventions: Drug: Prucalopride
- 5 (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- 4 (Active Comparator): Prucalopride
  Interventions: Drug: Prucalopride

INTERVENTIONS:
Drug: Prucalopride — 0.5 mg o.d.
  Other Names: Resolor
  Arms: 1
Other: Placebo — o.d.
  Arms: 5
Drug: Prucalopride — 1 mg o.d.
  Other Names: Resolor
  Arms: 2
Drug: Prucalopride — 2 mg o.d.
  Other Names: Resolor
  Arms: 3
Drug: Prucalopride — 4 mg o.d.
  Other Names: Resolor
  Arms: 4

SUMMARY:
The purpose of this study is to determine whether prucalopride is safe and effective in the treatment of constipation in elderly subjects living in a nursing facility.

Hypothesis:

Prucalopride up to a dose of 4 mg once daily is safe and well tolerated in in elderly subjects living in a nursing facility.

DETAILED DESCRIPTION:
This is a multicenter, Phase II, dose-escalation trial with a 4 week double-blind, placebo-controlled treatment period. There will be four treatment cohorts (0.5 mg, 1 mg, 2 mg, or 4 mg) with 25 subjects in each. The first cohort of 25 subjects will be randomly assigned to receive either 0.5 mg R108512 or placebo in a 4 to 1 ratio, respectively, for four weeks. After two weeks of treatment, the safety and tolerability of this dose will be evaluated for each subject by an independent (external) safety committee. If, at the completion of treatment, the safety committee grants approval to proceed to a higher dose, the second cohort will be randomly assigned to receive either 1 mg R108512 or placebo for four weeks. In a likewise manner, each dose will be evaluated for safety and tolerability before the next cohort will be treated with a higher dose. No subject can participate in more than one treatment cohort.

Subjects will be instructed not to change their diet or lifestyle during the trial. Subjects will be allowed to continue the use of routine stool softeners and fiber supplements during the trial; however, all existing stimulant or osmotic laxative medication will be withdrawn. If, during the trial, the subject does not have a complete bowel movement for three or more consecutive days, he/she will be allowed the use of his/her usual stimulant or osmotic laxative or an enema as a rescue medication. No laxatives or enemas should be used within the 24 hours before and 24 hours after the start of double-blind treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients at least 65 years of age (no upper age limit).
2. History of constipation. i.e., the patient should have received any treatment for constipation at any time during the 4 weeks (28 days) preceding entry into the study, including fibre/bulk forming supplements.
3. The patient had to live in a nursing facility.
4. The patient had to be clinically stable.
5. The patient had to be able to take oral medications.
6. The patient had to be continent of bowels the majority of time.
7. The patient had to be able to reliably communicate AEs.
8. The patient had to provide informed consent, signed by the patient or legally acceptable representative and by the investigator.

Exclusion Criteria:

1. Patients who were known to be HIV positive or who had AIDS.
2. Patients who were being actively treated with Propulsid (cisapride) or cancer chemotherapy other than hormonal agents.
3. Patients with significantly impaired renal function, i.e., creatinine clearance <30 mL/min using the Cockcroft and Gault formula:

   Males: CLCR = [(140-age) x (weight in kg)] / 72 x (SCR).

   Females: CLCR = male value x 0.85

   Because the calculated value for creatinine clearance could be artificially high when serum creatinine concentrations were very low, patients with a serum creatinine <0.5 mg/dL were excluded from the study.
4. Patients who received an investigational drug in the 30 days preceding the study.
5. Patients who had previously received either R093877 or R108512.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 1999-02; Primary Completion 2000-05 (Actual); Study Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Patient's Global Assessment of severity of constipation and efficacy of treatment evaluated (for exploratory reasons only). | 4 weeks

SECONDARY OUTCOMES:
Patient's symptom assessment(evaluated for exploratory reasons only). | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: D O'Neill, MD, Principal Investigator — Riverside Regional Convalescent Center

REFERENCES:
- [Derived] Camilleri M, Beyens G, Kerstens R, Robinson P, Vandeplassche L. Safety assessment of prucalopride in elderly patients with constipation: a double-blind, placebo-controlled study. Neurogastroenterol Motil. 2009 Dec;21(12):1256-e117. doi: 10.1111/j.1365-2982.2009.01398.x. Epub 2009 Sep 9. PMID 19751247